CLINICAL TRIAL: NCT03179228
Title: Phase II, Single Arm Prospective Study To Evaluate Safety And Efficacy Of Prostate Artery Embolization In Patients With Lower Urinary Tract Symptoms Due To Benign Prostatic Hyperplasia
Brief Title: Prostate Artery Embolization for the Treatment of Benign Prostatic Hyperplasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA approved Embospheres for prostate embolization, so IDE not needed
Sponsor: John D Louie (Other)
Responsible Party: Sponsor-Investigator, John D Louie, Clinical Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAE-01
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Prospective Single Center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prostate Embolization (Experimental): Prostate Embolization with acrylic polymer microspheres impregnated with porcine gelatin
  Interventions: Device: Prostate Embolization

INTERVENTIONS:
Device: Prostate Embolization — Embolization of the prostate with acrylic polymer microspheres impregnated with porcine gelatin

SUMMARY:
The primary study objective is to evaluate improvement of symptoms from benign prostatic hyperplasia (BPH) as assessed by the International Prostate Symptom Score (IPSS) at 12 months post prostatic artery embolization (PAE) with bland microspheres.

DETAILED DESCRIPTION:
This is a phase II, single center, prospective, single arm, investigational study to evaluate the safety and efficacy of prostate artery embolization (PAE) for treatment of severe lower urinary tract symptoms (LUTS) related to BPH in patients with prostate size greater than 40 grams that either refuse surgical treatment or are considered poor candidates for traditional surgical therapy. Two hundred patients will be enrolled in the single treatment arm with follow-up for no less than 12 months.

The study will involve a screening period in which patient eligibility will be determined. Once eligibility is confirmed, patients will receive PAE with bland microspheres within 4 weeks of screening baseline imaging. After treatment, patients will return for follow-up visits at 1 month, 3 months, 6 months, and 12 months post PAE. At each of these visits, patients will complete IPSS and IIEF questionnaires, undergo a physical exam, laboratory assessment (including PSA) and perform a medication review. Repeat TRUS and uroflowmetry will be performed at the 3, 6, and 12 month post PAE follow-up visits. MRI or CT will be conducted at the 3 and 12 month visit. Cystoscopy and proctoscopy will be performed if medically indicated.

The primary endpoint will be improvement of BPH symptoms as assessed by the IPSS at 12 months post PAE. Patients will continue to be followed according to the institutional standard of care follow-up schedule after they complete the study.

Safety will be evaluated throughout the initial 12 months of the study by assessing adverse events and findings on physical examination. Concomitant medication usage will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged 50 years or older.
2. Patient has signed informed consent
3. Patient has experienced lower urinary tract symptoms (LUTS) for at least 6 months prior to study enrollment
4. Patient has a prostate size larger than 40g as measured by MRI or CT (if MR not possible)
5. Patient has an IPSS score greater than or equal to 13
6. Patient either:

   i. Refuses surgical treatment ii. Is considered high risk for surgical treatment
7. Patient is either:

   i. Refractory to medical treatment ii. Contraindicated for medical treatment
8. Patient must meet ONE of the following criteria:

   * Baseline PSA ≤ 2.5ng/mL
   * Baseline PSA > 2.5 ng/mL and ≤ 10 ng/mL AND free PSA ≥ 25% of total PSA (no biopsy required)
   * Baseline PSA > 2.5 ng/mL and ≤ 10 ng/mL AND free PSA < 25% of total PSA AND negative prostate biopsy result (minimum of 12 core biopsy) within 12 months
   * Baseline PSA >10 ng/mL AND negative prostate biopsy result (minimum of 12 core biopsy) within 12 months
9. Patient has a peak urine flow rate < 12ml/sec.

Exclusion Criteria:

1. Active prostatitis or urinary tract infection
2. History of prostate or bladder cancer, or currently being evaluated for cancer
3. Bladder atonia, neurogenic bladder disorder or other neurological disorder that is impacting bladder function.
4. Urethral stricture, bladder neck contracture, other potentially confounding bladder pathology, bladder disease, or confounding urethral pathology
5. Patient has taken beta blockers, antihistamines, anticonvulsants, or antispasomodics within 1 week of study treatment AND has not been on the same drug dosage for 6 months with a stable voiding pattern.
6. Patient has taken antidepressant, anticholinergics, androgens or gonadotropin-releasing hormonal analogues within 2 months of study treatment AND has not been on the same drug dosage for at least 3 months with a stable voiding pattern.
7. Patient has taken alpha blockers within 4 weeks of study treatment AND has not been on the same drug dosage for at least 3 months with a stable voiding pattern.
8. Patient has taken 5-alpha reductase inhibitors within 3 months of study treatment AND has not been on the same drug for at least 6 months with a stable voiding pattern
9. History of open prostate surgery, radiofrequency, or microwave therapy
10. Previous open bladder or rectosigmoid colon surgery
11. Acute urinary retention requiring an indwelling catheter
12. Cystolithiasis within the past 3 months
13. Coagulation disturbances not normalized by medical treatment
14. Iodinated contrast allergy not controlled with 24-hour steroid preparation
15. History of pelvic irradiation
16. History of severe peripheral vascular disease or known major iliac arterial occlusive disease
17. Interest in future fertility
18. Significant cardiac or respiratory disease that the Investigator believes puts the patient at risk for a complication during the procedure
19. Acute urinary retention requiring an indwelling catheter
20. Life expectancy less than 6 months
21. History of rectal disease
22. Known immunosuppression either pathological or pharmacological
23. Presence of collateral vessel pathways potentially endangering normal anatomy during embolization that cannot be bypassed with the microcatheter
24. History of any illness or surgery that might confound the results of the study, by producing symptoms which may be confused with those of the disease process under consideration (e.g., Parkinson's, multiple Sclerosis), or which pose an additional risk to the patient.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-14 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate improvement of symptoms from benign prostatic hyperplasia | 12 months
  The primary study objective is to evaluate improvement of symptoms from benign prostatic hyperplasia (BPH) as assessed by the International Prostate Symptom Score (IPSS) in a whole number score.

SECONDARY OUTCOMES:
prostate specific antigen (PSA) | 12 months
  Change in ng/mL from baseline
prostate size | 12 months
  prostate size measured in grams, as determined by TRUS or MRI
peak urine flow rate (Qmax) | 12 months
  Change from baseline in as measured in ml/sec
post-void residual urine volume (PVR) | 12 months
  ml of urine in the bladder after urination
Erectile Function Survey | 12 months
  as measured in 5. Change from baseline in erectile function as assessed by the International Change from baseline in erectile function as assessed by the International Index of Erectile Function (IIEF) in whole numbers

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uflacker A, Haskal ZJ, Bilhim T, Patrie J, Huber T, Pisco JM. Meta-Analysis of Prostatic Artery Embolization for Benign Prostatic Hyperplasia. J Vasc Interv Radiol. 2016 Nov;27(11):1686-1697.e8. doi: 10.1016/j.jvir.2016.08.004. Epub 2016 Oct 12. PMID 27742235
- [Background] Carnevale FC, Iscaife A, Yoshinaga EM, Moreira AM, Antunes AA, Srougi M. Transurethral Resection of the Prostate (TURP) Versus Original and PErFecTED Prostate Artery Embolization (PAE) Due to Benign Prostatic Hyperplasia (BPH): Preliminary Results of a Single Center, Prospective, Urodynamic-Controlled Analysis. Cardiovasc Intervent Radiol. 2016 Jan;39(1):44-52. doi: 10.1007/s00270-015-1202-4. Epub 2015 Oct 27. PMID 26506952